CLINICAL TRIAL: NCT05895214
Title: MESOPANC-01 Study: The Mesopancreas and the Ductal Adenocarcinoma of the Pancreatic Head: From Preoperative Imaging to Histopathological and Surgical Outcome
Brief Title: Mesopancreas Study in Pancreatic Cancer
Acronym: MESOPANC-01
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: DRKS000295
Record Dates: First submitted 2023-04-25; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: PDAC; Pancreatoduodenectomy; Margin, Resection; Surgery; Local Recurrent Tumor
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who received primary surgery: preoperative CT scans available for assessing resectability criteria and presumed mesopancreatic infiltration status (CT scans are centrally evaluated) UICC 8th edition staging including CRM Tumor size in mm measured twice perpendicular Age Sex CA 19-9 values (preoperative) ECOG status BMI Type of PD (tail preserved vs total PD) simultaneous vessel resection (complete, partial; combined arterial and venous)
  Interventions: Procedure: oncological relevance of the mesopancreas
- patients who received neoadjuvant treatment prior to surgery: Peri-therapeutic CT scans available for assessing resectability criteria and presumed mesopancreatic infiltration status (CT scans are centrally evaluated) UICC 8th edition staging including CRM Tumor size in mm measured twice perpendicular Age Sex CA 19-9 values (peri-therapeutic) ECOG status BMI Type of neoadjuvant Therapy Type of PD (tail preserved vs total PD), simultaneous vessel resection (complete, partial; combined arterial and venous) Tumor response according to CAP
  Interventions: Procedure: oncological relevance of the mesopancreas

INTERVENTIONS:
Procedure: oncological relevance of the mesopancreas — Invasion status Invasion depth in mm Depth of mesopancreas in mm Treitz fascia intact (histopathological examination)

SUMMARY:
After the Introduction of the pathological circumferential resection margin (CRM status by LEEPP Protocol), residual cancer (R1 resection) was most often found in the dorsal and medial resection margins. Yet only the medial resection margin is preoperatively evaluated during staging, while the dorsal resection margin which embeds the mesopancreatic fat and thus resembles the area of the mesopancreas, is not considered during preoperative assessment for resectability. Local recurrence is similarly prevalent as systemic relapse, and revised lower rates of R0CRM- resections through the LEEPP protocol explained the poor local tumor control. The aim of this study is to interdisciplinary approach the circumferential infiltration status of the PDAC concentrating foremost on the mesopancreas of the dorsal resection margin by including anatomic and embryologic derived perspectives.

DETAILED DESCRIPTION:
For patients with a ductal adenocarcinoma of the pancreatic head (PDAC) pathological evaluation of the pancreatoduodenectomy specimen has endured a redefined process. After the Introduction of the pathological circumferential resection margin, residual cancer (R1 resection) was most often found in the dorsal and medial resection margins. Yet only the medial resection margin is preoperatively evaluated by staging and utilized during assessment of resectability. The dorsal resection margin which resides residual cancer (R1 resection) at a similar rate compared to the medial resection margin, is not considered during preoperative assessment for resectability. After the inclusion of the pathological LEEPP protocol true R0 resection rates have dropped to ~30%.

Next to the poor systemic tumor control and thus early detected relapse in PDAC patients, local recurrence is evenly at risk and remains an ungoing dilemma. Revised pathological outcome by the implemented LEEPP protocol explains the poor local tumor control.

The aim of this study is to interdisciplinary approach the circumferential infiltration status of the PDAC concentrating foremost on the dorsal resection margin by including anatomic and embryologic derived perspectives.

These perspectives have already been implemented by complete mesocolic and total mesorectal excision. The mesocolon of the ascending colon is embedded dorsally by fascia sheets, resulted by the embryologic fusion process, and the anatomic landmark of this fascia sheet has gained significant clinical relevance for radical surgical resection (Toldt fascia for total mesocolic excision). While surgical perspectives for the colorectal system have included the anatomic and embryologic nature of the colon and rectum, these landmarks and the idea of ''compartment anatomy'' are not implemented during pancreatoduodenectomy.

It seems rational to suggest that redefined surgical standards for colorectal cancer patients with implemented fascial sheets as anatomic landmarks could be translated to the pancreas as well. Similar to the ascending colon; the pancreas remains secondary retroperitoneal. The Treitz fascia is a cranio-medial extension of the toldts fascia, which again is an anatomic landmark for total mesocolic excision. The superior mesenteric artery serves as an anchor point for the embryologic rotation process of the pancreas until it remains secondary retroperitoneal. From an anatomic and embryologic point of view, there should not be any doubt for the existence of a mesopancreas.

The medial resection margin after pancreatoduodenectomy is resembled mostly by the portal confluens and does not embed any peripancreatic fat from the mesopancreas, underlining the different embryologic anlage between the pancreas and the portal venous system. The mesopancreas is located underneath the portal confluens, between the duodenum/pancreatic tissue and the inferior caval vein/abdominal aorta and continually encompasses the SMA. The dorsal resection margin during pancreatoduodenectomy resembles the mesopancreas and the aim of this multicentric prospective study is to study the oncological relevance of the mesopancreas.

Neoadjuvant therapy is a rising option for PDAC patients, and resectability criteria have been implemented to adequately stage these patients prior to therapy initiation. Current guidelines recommend to preoperatively investigate the medial vascular axis which represents the medial vascular groove. Patients are therefore sub-grouped into primary resectable, borderline resectable and non resectable mainly on the presumed infiltration status of the portomesenteric system.

In summary, the infiltration status of the PDAC is mainly being concentrated on the vascular groove. However, the dorsal resection margin, which is evenly at risk for incomplete resection (CRM assessment), is not considered during resectability stratification. Steps to secure or preoperatively assess this mesopancreatic area are not considered yet.

To stratify patients adequately for individualized therapy (neoadjuvant treatment vs surgery) a circumferential assessment, is crucial. Yet a circumferential assessment of the PDAC is provided only pathologically. In our opinion to realize a complete frame of tumor extensions a circumferential assessment should be implemented radiographically and surgically as well.

This observational study in patients with a ductal adenocarcinoma of the pancreatic head (PDAC) is of a prospective multicentric nature. In this study the mode of multimodal treatment, pre-operative computed tomographic staging, biological status (CA-19-9 values) are analyzed in a prospective consecutive treated patient cohort with respect to the infiltration status of the mesopancreas. The infiltration status of the mesopancreas is histopathologically analyzed while evaluating the dorsal resection margin for resection margin status (status positive/negative, depth of invasion in mm, depth of mesopancreas in mm, status of intact fascia sheet). No control group or placebo group exists.

The aim of this study is to analyze the oncological relevance of mesopancreatic fat infiltration both in upfront resected and neoadjuvant treated PDAC patients and to evaluate the feasibility of computed tomographic staging and preoperative serologic CA 19-9 values to predict the mesopancreatic infiltration status.

The histopathological analysis in each study center is an obligatory tool in order to postoperatively stage the PDAC. For this instance, the mesopancreatic fat infiltration status is analyzed in each respective study center. The radiographic analysis of the mesopancreas has yet not been standardized. For this mater, preoperative and peri-chemotherapeutic CT slides are centrally evaluated by the leading study initiators.

ELIGIBILITY:
Inclusion Criteria:

* All patients age ≥18 years who are admitted for primary surgery or patients who Received neoadjuvant therapy prior to surgery
* CRM analysis through Pathologic Institute in study centre already implemented (see LEEPP protocol Menon et al (2009) Impact of margin status on survival following pancreatoduodenectomy for cancer: the Leeds Pathology Protocol (LEEPP). HPB 11(1):18-24)
* Preoperative computed-tomographic Imaging (biphasic) prior to surgery (if resected without neoadjuvant treatment)
* Pre-chemotherapeutic computed-tomographic and post-chemotherapeutic computed-tomographic if neoadjuvantly treated (biphasic).
* indepth information of surgical procedure (pancreatic tail preserved:yes/no, pylorus preserved resection: yes/no, venous resection: complete/partial/no, arterial resection: complete/partial/no)

Exclusion Criteria:

* Palliation
* Abort of operative procedure
* No preoperative computed-tomography for staging
* No pathological CRM Implementation according to the LEEPP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive treated patients who are diagnosed with PDAC and received upfront surgical resection or neoadjuvant treatment prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of mesopancreatic infiltration in a multicentric setting. | through study completion, an average of 1 year
  Rate of mesopancreatic fat infiltration
Statistical comparison of the mesopancreatic infiltration status with known oncologically relevant histopathological staging factors: is there a more aggressive tumor biology or an unfavorable tumor topography | through study completion, an average of 1 year
  Status of MP infiltration (pathologically analysed) vs. UICC and AJCC staging system (questionnaire from pathological staging reporting)
Statistical comparison of mesopancreatic infiltration status with the CRM of the dorsal resection margin and with the entire CRM | through study completion, an average of 1 year
  Status of MP infiltration (pathologically analysed) vs. R-status (R0CRM- vs. R0CRM+/R1)(questionnaire from pathological staging reporting)
Prediction value of density analyses in computed tomography (Hounsfield Unit) with mesopancreatic infiltration status in primary and neoadjuvantly patients | through study completion, an average of 1 year
  Density score of mesopancreas (HU) vs. Infiltration status of MP (Hounsfield Unit scale resembles the density assessment during computed tomography)(Hypothesis: higher HU measurements indicate higher risk for mesopancreatic fat infiltration) (minimum HU value: air -1000HU, maximum HU value: gold +30000 HU)

SECONDARY OUTCOMES:
Rate of mesopancreatic infiltration in primary and borderline resectable pancreatic head carcinomas (classification of resectability using the well-known ABC scheme) | through study completion, an average of 1 year
  Status of MP infiltration vs. resectability status
Incidence rate of mesopancreatic infiltration between neoadjuvant treated and primary resected patients (matched-pairs analysis: both patient groups (neoadjuvant vs. primary resected) must have similar resectability criteria). | through study completion, an average of 1 year
  Status of MP infiltration vs. treatment protocol (matched pair analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Sami Alexander Safi, MD, Principal Investigator — Department of Surgery (A), University Hospital of Duesseldorf of the Heinrich Heine University Duesseldorf, Germany
Locations (1):
- University Hospital Duesseldorf, Heinrich Heine University, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Agreement between Sponsor and research sight

REFERENCES:
- [Background] Safi SA, Haeberle L, Fluegen G, Lehwald-Tywuschik N, Krieg A, Keitel V, Luedde T, Esposito I, Rehders A, Knoefel WT. Mesopancreatic excision for pancreatic ductal adenocarcinoma improves local disease control and survival. Pancreatology. 2021 Jun;21(4):787-795. doi: 10.1016/j.pan.2021.02.024. Epub 2021 Mar 17. PMID 33775563
- [Background] Safi SA, Haeberle L, Heuveldop S, Kroepil P, Fung S, Rehders A, Keitel V, Luedde T, Fuerst G, Esposito I, Ziayee F, Antoch G, Knoefel WT, Fluegen G. Pre-Operative MDCT Staging Predicts Mesopancreatic Fat Infiltration-A Novel Marker for Neoadjuvant Treatment? Cancers (Basel). 2021 Aug 28;13(17):4361. doi: 10.3390/cancers13174361. PMID 34503170
- [Background] Safi SA, Haeberle L, Rehders A, Fung S, Vaghiri S, Roderburg C, Luedde T, Ziayee F, Esposito I, Fluegen G, Knoefel WT. Neoadjuvant Treatment Lowers the Risk of Mesopancreatic Fat Infiltration and Local Recurrence in Patients with Pancreatic Cancer. Cancers (Basel). 2021 Dec 23;14(1):68. doi: 10.3390/cancers14010068. PMID 35008232
- [Background] Esposito I, Kleeff J, Bergmann F, Reiser C, Herpel E, Friess H, Schirmacher P, Buchler MW. Most pancreatic cancer resections are R1 resections. Ann Surg Oncol. 2008 Jun;15(6):1651-60. doi: 10.1245/s10434-008-9839-8. Epub 2008 Mar 20. PMID 18351300
- [Background] Menon KV, Gomez D, Smith AM, Anthoney A, Verbeke CS. Impact of margin status on survival following pancreatoduodenectomy for cancer: the Leeds Pathology Protocol (LEEPP). HPB (Oxford). 2009 Feb;11(1):18-24. doi: 10.1111/j.1477-2574.2008.00013.x. PMID 19590619